CLINICAL TRIAL: NCT00619021
Title: A Phase I Study Evaluating Bronchial Artery Infusion (BAI) of Gemcitabine in Recurrent or Progressive Non-Small Cell Lung Cancer
Brief Title: Bronchial Artery Infusion of Gemcitabine in Treating Patients With Recurrent or Progressive Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding and study drugs unavailable
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002LS028; UMN-IRB-0201M15401 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-02-19; First posted 2008-02-20 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): Patient receives gemcitabine 600 mg/m^2.
  Interventions: Drug: gemcitabine hydrochloride
- Cohort 2 (Experimental): Patient receives gemcitabine 800 mg/m^2.
  Interventions: Drug: gemcitabine hydrochloride
- Cohort 3 (Experimental): Patient receives gemcitabine 1000 mg/m^2.
  Interventions: Drug: gemcitabine hydrochloride
- Cohort 4 (Experimental): Patient receives gemcitabine 1200 mg/m^2.
  Interventions: Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride — 4 dose levels designated by cohort; 600 mg/m^2, 800 mg/m^2, 1000 mg/m^2, 1200 mg/m^2
  Other Names: Gemzar

SUMMARY:
RATIONALE: Bronchial artery infusion uses a catheter to deliver antitumor substances directly to the lungs. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving gemcitabine in different ways may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of gemcitabine given by bronchial artery infusion and to see how well it works in treating patients with recurrent or progressive non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the maximum tolerated dose of gemcitabine hydrochloride delivered via bronchial artery infusion in patients with recurrent or progressive non-small cell lung cancer.

Secondary

* To evaluate local response in patients treated with this therapy.
* To characterize the pharmacokinetics of gemcitabine hydrochloride in patients treated with this therapy.

OUTLINE: This is a dose-escalation study of gemcitabine hydrochloride delivered via bronchial artery infusion.

Patients receive gemcitabine hydrochloride via bronchial artery infusion over 30-60 minutes on day 1 and via IV infusion over 30 minutes on day 8 of course 1. Patients then receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 of all subsequent courses. Treatment repeats every 21 days in the absence of disease progression and unacceptable toxicity.

After completion of study therapy, patients are followed every 8 weeks to 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed non-small cell lung cancer meeting the following criteria:

  * No T2 lesions invading the visceral pleura, causing atelectasis, or proximal to an obstructing pneumonia
  * No T3 lesions invading the chest wall (including the parietal pleura, musculature, and/or rib), mediastinal pleura, diaphragm, or pericardium
  * No T4 lesions invading the heart, great vessels, carina, or esophagus
* Must have disease that is incurable by standard treatment, defined as a minimum of first-line therapy with a platinum-containing regimen and second-line therapy with docetaxel, pemetrexed disodium, or erlotinib hydrochloride
* Measurable or nonmeasurable disease as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Serum creatinine ≤ 3.0 mg/dL
* Total bilirubin < 1.5 times upper limit of normal
* International normalized ratio (INR) ≤ 1.3
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective non-hormonal contraception

Exclusion Criteria:

* Superior vena cava syndrome or superior sulcus tumors
* Patients with airway obstructing lesions, or patients experiencing hemoptysis, dyspnea, chest pain, and/or copious sputum production may be eligible after careful consideration by the study physicians
* Prior or concurrent malignancy except inactive nonmelanoma skin cancer, carcinoma in situ of the cervix, stage I carcinoma of the prostate with normal PSA, or other cancer from which the patient has been disease free for 3 years
* Medical conditions that would make this protocol unreasonably hazardous, in the opinion of the treating physician, including any of the following:

  * Uncontrolled infection (including HIV)
  * Poorly controlled diabetes mellitus
  * Active cardiac disease (i.e., unstable angina, myocardial infarction within the past 6 months, or congestive heart failure)
* Other serious medical illness that would limit survival to < 3 months, or psychiatric condition that would prevent informed consent, unless a legal guardian is available
* Must consent to participate in the laboratory study, "Population Pharmacokinetics and Pharmacogenetics of Gemcitabine in Adult Patients with Solid Tumors" during course 1
* More than 6 months since prior gemcitabine hydrochloride

  * More than 2 weeks since other prior chemotherapy
* More than 4 weeks since prior radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and dose-limiting toxicity of gemcitabine hydrochloride when administered via bronchial artery infusion | At time of dose-limiting toxicity

SECONDARY OUTCOMES:
Local response as measured by RECIST | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D'Cunha, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States